CLINICAL TRIAL: NCT01190020
Title: Effect of Lubiprostone on Methanogenesis and Bowel Function in Chronic Constipation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Principal Investigator, Satish Rao, PI, University of Iowa
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: MS-LUB-106
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2018-07

CONDITIONS: Chronic Constipation, Methanogenesis
MeSH Terms: interventions — Lubiprostone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lubiprostone (Active Comparator): 24mcg BID for 4 weeks, oral medication
  Interventions: Drug: Lubiprostone
- Placebo (Placebo Comparator): 24mcg BID for 4 weeks (placebo), oral medication
  Interventions: Drug: Lubiprostone Control

INTERVENTIONS:
Drug: Lubiprostone — Colonic transit study performed and stool/symptom diaries will be reviewed. Eligible subjects will be given a lactulose breath test and randomized to Lubiprostone or placebo. Treatment group receives 24 mcg Lubiprostone twice daily and placebo group receives pills (identical in appearance to the study drug) for one month. Subjects will be asked to maintain a daily stool/symptom diary for duration of the study. In the middle of the study a research coordinator will call the subjects to take questions/concerns and record adverse events. Lactulose breath test will be repeated, constipation questionnaire filled out, colon transit study performed.
  Arms: Lubiprostone
Drug: Lubiprostone Control — Colonic transit study performed and stool/symptom diaries will be reviewed. Eligible subjects will be given a lactulose breath test and randomized to Lubiprostone or placebo. Treatment group receives 24 mcg Lubiprostone twice daily and placebo group receives pills (identical in appearance to the study drug) for one month. Subjects will be asked to maintain a daily stool/symptom diary for duration of the study. In the middle of the study a research coordinator will call the subjects to take questions/concerns and record adverse events. Lactulose breath test will be repeated, constipation questionnaire filled out, colon transit study performed.
  Arms: Placebo

SUMMARY:
Lubiprostone, a chloride channel activator, has been shown to improve symptoms of chronic constipation, largely by enhancing chloride-rich intestinal fluid secretion. Whether Lubiprostone has effects on colonic methanogenesis is not known. The investigators hypothesize that the effects of Lubiprostone may in part be due to its effects on altering colonic flora, particularly methanogenic flora.

By altering the colonic stasis of stool and through more efficient clearance of digestive residue, the investigators anticipate that Lubiprostone may either inhibit or promote better excretion of methanogenic flora, and thereby decrease the gut load of methane producing bacteria. In turn, this may lead to enhanced colonic smooth muscle contraction and an increased rate of spontaneous bowel movements and reduction of constipation symptoms.

The aim is to investigate the effects of Lubiprostone on intestinal methane production and bowel symptoms in patients with chronic constipation, by performing a randomized, double blind, placebo controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Constipation as defined by Rome III criteria13. Patients must have symptoms > 3 days/month for the past three months and report at least two of the following symptoms ≥ 25% of the time: straining, lumpy or hard stool, sensation of incomplete evacuation, sensation of anorectal obstruction/blockage, use of manual maneuvers, < 3 bowel movements/week. Also,they should have insufficient criteria for IBS, and only rarely loose stools without the use of laxatives.
* ≥ 3 ppm methane value at baseline1, 2(before sugar load).

Exclusion Criteria:

* Patients taking drugs that are known to be constipating will be excluded or asked to discontinue medications for at least 2 weeks and reassessed. For example, we will recommend that patients taking calcium channel antagonists contact their respective primary care physicians to explore alternative medications for hypertension such as beta blockers or ACE-inhibitors. If the calcium channel antagonists are able to be discontinued, patients will be re-screened at least two weeks after the medications are discontinued. If patients no longer meet inclusion criteria, they will be excluded from the study. Patients who remain constipated will be eligible for enrollment.
* Patients with co-morbid illnesses such as severe cardiovascular disease, chronic renal failure, or those with previous gastrointestinal surgery except cholecystectomy and appendectomy
* Patients with neurologic diseases such as multiple sclerosis, strokes, spinal cord injuries, and those who have problems with cognizance, i.e. a mini-mental score of <15 and/or are legally blind will be excluded.
* Women who are pregnant or are likely to conceive during the course of the study will be excluded. Urinary pregnancy tests will be performed on all women of child-bearing potential prior to enrollment and before any x-ray of the abdomen.
* Patients with Hirschsprung' s disease, or active local anorectal problems such as anal fissures, bleeding hemorrhoids, Crohn's, colitis, or colon cancer.
* Patients with alternating constipation and diarrhea and those who fulfill the Rome-III criteria for irritable bowel syndrome.
* Recent antibiotic use (last 6 weeks).
* Patients using laxatives, PEG or Tegaserod and unwilling to discontinue these medications at least 2 weeks prior to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Lubiprostone: Received 24 mcg of lubiprostone twice a day with meals.
- Placebo: Received placebo twice a day with meals.
Period: Overall Study
Arm/Group | Lubiprostone | Placebo
Started | 29 | 12
Completed | 22 | 12
Not Completed | 7 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lubiprostone | Placebo | Total
Number analyzed (Participants) | 29 | 12 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 11 | 37
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (11.9) | 47.3 (22.5) | 43.7 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 12 | 37
  Male | 4 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 29 | 12 | 41

OUTCOME MEASURES:

1. Primary Outcome: Change in Methane Production
Description: Change in the mean area under the curve of the breath hydrogen and methane gas profiles in parts per million, from time 0 to 120 minutes, between baseline versus mean area under the curve at the end of study.
Time Frame: Baseline and 1 month
Population: patients who completed the study were analyzed
Measure: Mean (Standard Error); unit: parts per million*minutes
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 22 | 12
parts per million*minutes | 10645 (1481) | 14635 (2330)

2. Secondary Outcome: Stool Frequency (Complete Spontaneous Bowel Movements)
Description: change in mean stool frequency (delta) between baseline week and final week of study
Time Frame: Baseline and 1 month
Population: subjects who completed the study
Measure: Mean (Standard Error); unit: bowel movements per week
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 22 | 12
bowel movements per week | 3.71 (0.84) | 0.85 (0.54)

3. Secondary Outcome: Percentage Change in the Colonic Transit Time
Description: Percentage change of colonic transit time between the baseline colonic transit study and the colonic transit study at the end of study
Time Frame: Baseline and 1 month
Population: subjects who completed the study
Measure: Mean (Standard Error); unit: percent
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 22 | 12
percent | 0.23 (0.06) | 0.48 (0.1)

4. Secondary Outcome: Peak Methane Value
Description: The peak methane value measured during the baseline breath study will be compared with the peak methane obtained at the end of study breath test
Time Frame: Baseline and 1 month
Measure: Mean (Standard Error); unit: parts per million
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 22 | 12
parts per million | 51.3 (7.1) | 70.5 (11.2)

ADVERSE EVENTS:
Arm/Group | Lubiprostone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/12
Other Adverse Events (participants affected / at risk) | 4/29 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lubiprostone (N=29) | Placebo (N=12)
Chest Tightness (Respiratory, thoracic and mediastinal disorders) | 2 | 0 — 2 subjects experience chest tightness and shortness of breath within one hour of taking the pill.
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2 | 0 — 2 subjects experienced chest tightness and shortness of breath within one hour of taking the pill.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No